CLINICAL TRIAL: NCT06186063
Title: The Role of Amylin in Bone Metabolism
Acronym: AmyBone
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Filip Krag Knop (Other)
Responsible Party: Sponsor-Investigator, Filip Krag Knop, Professor, MD, PhD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-22050946
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Bone Diseases, Metabolic; Type 1 Diabetes
MeSH Terms: conditions — Bone Diseases, Metabolic; Diabetes Mellitus, Type 1 | interventions — pramlintide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The investigators apply a randomized, double-blinded, placebo-controlled, crossover design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pramlintide infusion (Experimental): A stable amylin analogue.
  Interventions: Other: Pramlintide
- Placebo infusion (Placebo Comparator): Isotonic saline (0.9% NaCl).
  Interventions: Other: Placebo (saline) infusion

INTERVENTIONS:
Other: Pramlintide — At time 0 min, continuous infusion of a stable amylin analogue (pramlintide) will be initiated at a rate of 3.0 pmol/kg/min. The infusion will be terminated after 180 minutes.
  Arms: Pramlintide infusion
Other: Placebo (saline) infusion — At time 0 min, continuous infusion of isotonic saline will be initiated at a rate of 150 ml/h. The infusion will be terminated after 180 minutes.
  Arms: Placebo infusion

SUMMARY:
The clinical study aims to investigate the effect of the intravenously administrated amylin analogue (pramlintide) on the circulating levels of C-terminal telopeptide of type I collagen (CTX-1) (a marker of bone resorption) and N-terminal propeptide of type I procollagen (P1NP) (a marker of bone formation) in individuals with type 1 diabetes and matched healthy controls during fasting euglycemic conditions.

DETAILED DESCRIPTION:
Using a randomised double blinded placebo-controlled crossover design the investigators will evaluate the effects of the intravenously administrated amylin analogue (pramlintide) on circulating levels of CTX-1 and P1NP in ten individuals with type 1 diabetes and ten healthy controls matched for age, gender and body mass index (BMI) during fasting and euglycemic conditions. Each participant will receive double-blinded infusions of pramlintide (3 pmol/kg/min) and saline on two separate study days performed in randomised order.

The primary endpoints are the relative changes in the plasma levels of P1NP and CTX-1. The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma CTX-1 and P1NP as well as %-changes from baseline including nadir.

The secondary endpoints encompass changes in plasma concentrations of calcium, parathyroid hormone (PTH), alkaline phosphatase, osteocalcin, glucagon, insulin, C-peptide, glucose, glucose-dependent insulinotropic polypeptide and glucagon-like peptide 1 and glucagon-like peptide 2.

ELIGIBILITY:
Inclusion criteria type 1 diabetes:

* Caucasian ethnicity
* Age between 18 and 60 years
* BMI between 18.5 and 27 kg/m2
* Type 1 diabetes (diagnosed according to the criteria of the World Health Organization) with HbA1c <69 mmol/mol (<8.5%) and
* Type 1 diabetes duration of 2-20 years
* C-peptide negative (stimulated C-peptide ≤30 pmol/l)
* Treatment with a stable basal-bolus or insulin pump regimen for ≥3 months
* Normal vitamin D (>50 nmol/l)
* Informed consent

Exclusion criteria type 1 diabetes:

* Anaemia (haemoglobin below normal range)
* Liver disease (ALAT and/or ASAT >2 times normal values) or history of hepatobiliary disorder
* Nephropathy (eGFR <60 ml/min/1,73m2 and/or microalbuminuria)
* Microvascular complications except non-proliferative retinopathy
* Treatment with anti-osteoporosis medication or glucocorticoids
* Fractures within the last 6 months
* For women: currently perimenopausal or postmenopausal
* Diseases affecting calcium metabolism (e.g. hypoparathyroidism, hyperparathyroidism, osteoporosis, vitamin D deficiency and cancer)
* Pregnancy or breastfeeding
* Any physical or psychological condition that the investigator feels would interfere with trial participation
* Treatment with any glucose-lowering drugs beside insulin, treatment with medication against osteoporosis or treatment with any form of glucocorticoids

Inclusion criteria healthy controls:

* Caucasian ethnicity
* Age between 18 and 60 years
* BMI between 18.5 and 27 kg/m2
* Fasting plasma glucose ≤7.0 mmol/l and glycated haemoglobin (HbA1c) <48 mmol/mol
* Normal blood haemoglobin (8.3-10.5 mmol/l (males) and 7.3 - 9.5 mmol/l (females))
* Normal plasma vitamin D (>50 nmol/l)
* Informed consent

Exclusion criteria healthy controls:

* Any form of diabetes (according to World Health Organization criteria)
* Anaemia (haemoglobin below normal range)
* Nephropathy (eGFR <60 ml/min/1,73m2 and/or microalbuminuria)
* Known liver disease and/or alanine transaminase (ALAT) or aspartate transaminase (ASAT) >2 × upper normal limit
* Any fractures within the last 6 months
* For women: currently perimenopausal or postmenopausal
* Diseases affecting calcium metabolism (e.g. hypoparathyroidism, hyperparathyroidism, osteoporosis, vitamin D deficiency and cancer)
* Pregnancy or breastfeeding
* Any condition considered incompatible with participation by the investigators

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Relative changes in the plasma levels of C-terminal telopeptide of type I collagen (CTX-1) | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma CTX-1 as well as %-changes from baseline including nadir.
Relative changes in the plasma levels of N-terminal propeptide of type I procollagen (P1NP) | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma P1NP as well as %-changes from baseline including nadir.

SECONDARY OUTCOMES:
Changes in plasma concentrations of glucagon. | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma levels as well as %-changes from baseline including nadir.
Changes in plasma concentrations of insulin. | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma levels as well as %-changes from baseline including nadir.
Changes in plasma concentrations of C-peptide. | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma levels as well as %-changes from baseline including nadir.
Changes in plasma concentrations of glucose. | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma levels as well as %-changes from baseline including nadir.
Changes in plasma concentrations of glucose-dependent insulinotropic polypeptide (GIP). | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma levels as well as %-changes from baseline including nadir.
Changes in plasma concentrations of glucagon-like peptide 1 (GLP-1). | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma levels as well as %-changes from baseline including nadir.
Changes in plasma concentrations of glucagon-like peptide 2 (GLP-2). | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma levels as well as %-changes from baseline including nadir.
Changes in plasma concentrations of calcium. | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma levels as well as %-changes from baseline including nadir.
Changes in plasma concentrations of parathyroid hormone (PTH) | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma levels as well as %-changes from baseline including nadir.
Changes in plasma concentrations of alkaline phosphatase | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma levels as well as %-changes from baseline including nadir.
Changes in plasma concentrations of osteocalcin | From -15 minutes to 180 minutes
  The changes in plasma concentrations will be assessed by the total and incremental (baseline-subtracted) area under the curve for plasma levels as well as %-changes from baseline including nadir.

CONTACTS AND LOCATIONS:
Overall Officials: Filip K. Knop, Professor, MD, PhD, Principal Investigator — Center for Clinical Metabolic Research, Gentofte Hospital, Denmark
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Capital Region, Denmark